CLINICAL TRIAL: NCT03273985
Title: Effectiveness of Deep Dry Needling in Subjects With Shortened Triceps Surae Originated by Myofascial Pain Syndrome
Brief Title: Effectiveness of Dry Needling in Shortened Triceps Surae Muscle
Acronym: DN-TS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de León (Other)
Collaborators: Universidad Complutense de Madrid (Other)
Responsible Party: Principal Investigator, César Calvo Lobo, Professor, PhD, MSc, PT, Universidad de León
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DN-TS-UCM
Record Dates: First submitted 2017-09-01; First posted 2017-09-06 (Actual); Last update posted 2017-12-08 (Actual); Status verified 2017-12

CONDITIONS: Trigger Point Pain, Myofascial; Myofascial Pain Syndrome
MeSH Terms: conditions — Myofascial Pain Syndromes | interventions — Dry Needling; Acupressure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry needling (Experimental)
  Interventions: Other: Dry needling
- Ischemic compression (Experimental)
  Interventions: Other: Ischemic compression

INTERVENTIONS:
Other: Dry needling — Trigger point deep dry needling
  Arms: Dry needling
Other: Ischemic compression — Trigger point ischemic compression
  Arms: Ischemic compression

SUMMARY:
To date, there are not studies about the effectiveness of dry needling versus ischemic compression in the triceps surae trigger points. A randomized clinical trial is carried out. A sample of 30 subjects are recruited and allocated into dry needling (n = 15) and ischemic compression (n = 15). Outcome measurements such as dorsal flexion range of motion, plantar pressures, temperature, superficial muscle activity and trigger points pressure pain threshold are measured immediately before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Myofascial pain syndrome in the triceps surae muscle, limitation of ankle dorsal flexion range of motion.

Exclusion Criteria:

* Neurologic disorders, pharmacologic treatment (within the previous 3 months), cognitive impairment, prosthesis in the lower limb, systemic or infectious diseases, autoimmune diseases, fibromyalgia, hypothyroidism, anticoagulants or antiplatelet agents, and fear of needles.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2017-12-06 (Actual); Study Completion 2017-12-06 (Actual)

PRIMARY OUTCOMES:
Range of motion | Change from Baseline Range of motion at 25 minutes
  Ankle dorsal flexion by means of the goniometer

SECONDARY OUTCOMES:
Plantar pressures | Change from Baseline Plantar pressures at 25 minutes
  Plantar pressures platform
Temperature | Change from Baseline Temperature at 25 minutes
  Thermal imaging
Superficial muscle activity | Change from Baseline Superficial muscle activity at 25 minutes
  Electromyography
Pressure pain threshold | Change from Baseline Pressure pain threshold at 25 minutes
  Algometer

CONTACTS AND LOCATIONS:
Locations (1):
- Fisiofuenla, Fuenlabrada, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Benito-de-Pedro M, Becerro-de-Bengoa-Vallejo R, Elena Losa-Iglesias M, Rodriguez-Sanz D, Lopez-Lopez D, Palomo-Lopez P, Mazoteras-Pardo V, Calvo-Lobo AC. Effectiveness of Deep Dry Needling vs Ischemic Compression in the Latent Myofascial Trigger Points of the Shortened Triceps Surae from Triathletes on Ankle Dorsiflexion, Dynamic, and Static Plantar Pressure Distribution: A Clinical Trial. Pain Med. 2020 Feb 1;21(2):e172-e181. doi: 10.1093/pm/pnz222. PMID 31502640